CLINICAL TRIAL: NCT05759728
Title: A Phase 1/2a, Multicenter, Open-Label, Dose Escalation and Expansion Study of CNA3103 (LGR5-targeted, Autologous CAR-T Cells) Administered to Adult Subjects With Metastatic Colorectal Cancer
Brief Title: A Study of CNA3103 (LGR5-targeted, Autologous CAR-T Cells) Administered to Subjects With Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Carina Biotech Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CNA3103-001
Record Dates: First submitted 2023-02-13; First posted 2023-03-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer Metastatic
Keywords: CAR-T; LGR5

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CNA3103 Monotherapy (Experimental): Single intravenous dose of CNA3103 at Day 0
  Interventions: Biological: CNA3103: 5 x 10^7 cells; Biological: CNA3103: 1.5 x 10^8 cells; Biological: CNA3103: 4.5 x 10^8 cells; Biological: CNA3103: 1.5 x 10^9 cells; Biological: CNA3103: 2.5 x 10^7 cells; Biological: CNA3103: 6.75 × 10^8 cells

INTERVENTIONS:
Biological: CNA3103: 5 x 10^7 cells — CNA3103: 5 x 10^7 cells - intravenous infusion
Biological: CNA3103: 1.5 x 10^8 cells — CNA3103: 1.5 x 10^8 cells - intravenous infusion
Biological: CNA3103: 4.5 x 10^8 cells — CNA3103: 4.5 x 10^8 cells - intravenous infusion
Biological: CNA3103: 1.5 x 10^9 cells — CNA3103: 1.5 x 10^9 cells - intravenous infusion
Biological: CNA3103: 2.5 x 10^7 cells — CNA3103: 2.5 x 10^7 cells - intravenous infusion
Biological: CNA3103: 6.75 × 10^8 cells — CNA3103: 6.75 × 10^8 cells - intravenous infusion

SUMMARY:
This study aims to determine the safety and best response of treatment with CNA3103 (Leucine-rich repeat-containing G protein-coupled receptor 5 [LGR5]-targeted, Autologous Chimeric Antigen Receptor (CAR) -T Cells), for participants with Metastatic Colorectal Cancer.

Participants may undergo a pre-screening biopsy procedure to determine expression of LGR5.

Participants will undergo screening procedures, including leukapheresis (collection of T cells) and lymphodepletion (chemotherapy), up to 47 days prior to CNA3103 dosing.

Participants will receive a single Intravenous dose of CNA3103.

Expansion cohorts will open after determination of the maximum tolerated dose and recommended phase 2 dose in the dose escalation stage.

Participants will be followed up, monitored and will attend study visits for safety and research related tests and procedures for 2 years until disease progression, unacceptable toxicity or intolerable adverse event/s, death or withdrawal of consent.

DETAILED DESCRIPTION:
This is a Phase 1/2a, multicenter, open-label study in adult subjects with metastatic colorectal cancer. (CRC). The study will consist of 2 segments:

Phase 1 Segment (Dose Escalation): a Bayesian Optimal Interval (BOIN) study design will be used to minimize any risks of exposure to the novel CNA3103 CAR-T cells during dose escalation while determining the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D). A minimum of 3 subjects per cohort will be enrolled at each dose level, with appropriate staggering of subjects within and between dose levels.

Phase 2a Segment (Dose Expansion): After determination of the MTD/RP2D, additional subjects will be enrolled and treated with CNA3103 at that dose to further assess the safety, PK, pharmacodynamic, and anti-tumor properties of CNA3103. Based upon safety data of these additional subjects, the Sponsor, in consult with the Investigators, may choose to enroll additional subjects at the same or a different dose.

ELIGIBILITY:
Inclusion Criteria:

* Signed written Informed Consent.
* Male and female subjects aged greater than or equal to18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Score 0 to 1.
* Histologically or cytologically confirmed metastatic colorectal cancer previously treated with no more than 2 prior fluoropyrimidine, oxaliplatin, and/or irinotecan-based regimens for metastatic disease. Antibody-drug conjugates (ADCs) administered in the metastatic setting are also considered cytotoxic treatment and would count as a prior regimen. Neoadjuvant/adjuvant treatment of resectable oligometastatic disease, does not count as a prior line of therapy in the palliative setting unless there is development of an unresectable local or distant recurrence within 6 months of its last dose.

Subjects who discontinue their prior regimen due to toxicity (in the absence of disease recurrence/progression) will also have their prior therapy count as one prior regimen. Anti-Kirsten rat sarcoma virus (Anti-KRAS) agents are also allowable. The planned lymphodepletion start date must be at least 4 weeks from last chemotherapy, biologic, radiotherapy, or investigational therapy (excluding bridging therapy), with resolution of all lingering toxicities to Grade ≤ 1, with the exception of neuropathy and alopecia.

Subjects previously treated in the adjuvant/neoadjuvant setting with an oxaliplatin/irinotecan regimen, who develop an unresectable local recurrence and/or metastatic disease within 6 months of the date of last oxaliplatin/irinotecan chemotherapy will have their adjuvant/ neoadjuvant therapy count as one prior regimen.

* Positive for any level of LGR5 expression in tumor biopsies.
* Measurable or evaluable disease per RECIST version 1.1. Subjects with lung metastases involving less than or equal to 20% of both lung fields and with good respiratory reserves would be deemed eligible as long as the lesions do not compromise airways, vascular, pleural, or mediastinal spaces. Both measurable and non-measurable (evaluable) lesions would count for this assessment.

Subjects whose lung metastases involve more than 20% of both lung fields should be discussed with the Sponsor in more detail, taking into account disease tempo, clinical symptoms, respiratory function and compromise (current or impending) of airways, vascular, pleural, or mediastinal spaces. Both measurable and non-measurable (evaluable) lesions would count for this assessment.

* Life expectancy of at least >12 weeks.
* Normal organ and marrow function.
* No clinically significant abnormalities in urinalysis results at Screening.
* No known clinically significant gastrointestinal disease within 28 days prior to enrolment.
* No ongoing requirement for anti-diarrheal therapy.
* For female subjects of childbearing potential and male subjects with partners of childbearing potential, agreement (by subject and/or partner) to use a highly effective form of contraception and to continue its use for 6 months after the last dose of IP.
* Women of childbearing potential must have a negative serum pregnancy test within 72 hours prior to CNA3103 administration.

Exclusion Criteria:

* Inability to comply with study and follow-up procedures.
* Women who are pregnant or lactating.
* Has BRAF-mutated colorectal cancer.
* Has received trifluridine/tipiracil (TAS-102) or regorafenib for metastatic disease.
* Treatment with chemotherapy, hormonal therapy, immunotherapy, biologic therapy, or radiation therapy as cancer therapy (excluding bridging therapy) within 4 weeks prior to the lymphodepletion start date.
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent in the previous 28 days prior to enrolment.
* Have received antibody-based therapies within the previous 28 days or 5 half-lives of the agent, whichever is shorter.
* Major surgery, in the previous 4 weeks prior to enrolment.
* Clinically detectable pleural effusion requiring drainage in the 4 weeks prior to enrolment.
* Any uncontrolled medical or psychiatric risk factors which would contraindicate the use or impair the ability of the subject to provide informed consent, receive protocol therapy or may impose excessive risk to the subject.
* Known central nervous system (CNS) disease.
* Current use of medications that may have the potential of QTc prolongation.
* Uncontrolled bacterial, viral, or fungal infection, requiring systemic therapy.
* Has a known infection with human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C, alcoholic or other hepatitis, or cirrhosis.
* Inability to be venipunctured and/or tolerate venous access.
* Second malignancies within 5 years prior to enrollment, except for those with a negligible risk of metastasis or death, such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent.
* Active autoimmune disease that is not controlled by non-steroidal anti-inflammatory drugs (NSAIDs), inhaled corticosteroids, or the equivalent of ≤10 mg/day prednisone.
* History of inflammatory bowel disease (active or past) or active peptic ulcer disease.
* History of connective tissue disorders.
* History of chronic leukemias.
* History of previous, whole abdomen radiation therapy (or total pelvic radiation therapy) or more than Grade 1 residual toxicity from previous radiation therapy.
* High cardiovascular risk, including, but not limited to, recent coronary stenting or myocardial infarction in the past year
* Left ventricular ejection fraction <50%.
* Have had a venous thromboembolic event requiring anticoagulation.
* Congenital or acquired long QT syndrome.
* QTc prolongation.
* History of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies.
* Patients with ascites, previous drainage of ascites, peritoneal caking, and/or significant peritoneal deposits at Baseline are excluded from participation in the study
* Patients with reduced liver reserves and/or possibility of hepatobiliary complications, including, but not limited to; portal hypertension, liver resection (segmentectomy, metastasectomy) in the previous 6 months, patients with existing biliary stents or the need to receive a biliary stent to relieve bile duct obstruction of any etiology, patients with cholelithiasis, patients who abuse alcohol or paracetamol (with or without concomitant alcohol abuse), patients who use herbal medicines, and patients with substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of treatment with CNA3103. | 24 Months
  Incidence of Treatment-Emergent Adverse Events
To determine the overall best response to CNA3103. | 24 Months
  Best response per Response Evaluation Criteria in Solid Tumors (RECIST).

SECONDARY OUTCOMES:
To determine the recommended Phase 2a dose (RP2D) of CNA3103 | 28 days
  Determined by dose limiting toxicities (DLTs)
To monitor for replication competent viral construct in blood specimens | 24 Months
  Viral construct presence will be monitored
To determine the Pharmacokinetics of CNA3103 | 24 Months
  Levels of CNA3103 cells measured
To determine overall survival | 24 Months
  Survival will be calculated from the onset of CNA3103 therapy.
Failure to treat | 8 Weeks
  Caused by manufacturing issues or patient related issues.
To determine progression-free survival | 24 months
  Calculated from the onset of therapy to disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Carina Biotech Investigators, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No